CLINICAL TRIAL: NCT06230016
Title: Evaluation of the Adhesion of Children and Adolescents Treated for Cancer to Personalized Support in Adapted Physical Activity
Brief Title: Adhesion of Children and Adolescents Treated for Cancer to Personalized Support in Adapted Physical Activity Program
Acronym: APADHOP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Grenoble (Other)
Collaborators: University Grenoble Alps (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-A02343-42
Record Dates: First submitted 2023-12-26; First posted 2024-01-29 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2023-12

CONDITIONS: Childhood Cancer; Adapted Physical Activity
Keywords: motivation; restraint
MeSH Terms: conditions — Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: questionnaires — human and social science questionnaire (specifically designed by the expert lab of Grenoble) on motivation and restraint perceived by patient and parents, elaborated especially for this study.
  Questionnaire administred before the start of current care APA programm and after 4 to 6 months.
Other: PedsQL quality of life questionnaires — validated PedsQL (The Pediatric Quality of Life Inventory) questionnaires administred to children (if adequate) and parents before the start of current care APA programm and after 4 to 6 months

SUMMARY:
Adapted physical activity session with a formed professional is proposed in standard care since 2022 in the immuno-hematological service to all children with newly diagnosed cancer or relapse.

The aim of this study is to keep the children in the APA programm during all the treatment lenght.

This study aims to evaluate by questionnaires the motivation keys and restraint from children and parents before the APA program starts (at diagnosis or relapse if not previously participating to an APA programm) and after 4 to 6 months of APA programm.

The final expected fallout is to enhance children adhesion to long term APA program by implementing tools in current practice to overcome restraints from young patients and their parents

DETAILED DESCRIPTION:
The literature and the French Cancer Plan confirm the benefits of physical activity for cancer patients, and underline the importance of developing appropriate physical activity support for children and adolescents, given their specific needs and the societal and public health challenge represented by these budding patients.

Despite the abundance of studies relating to physical activity in oncology, few data are available, particularly in the pediatric and adolescent/young adult population :

* on physical activity interventions initiated early and sustained over time
* on personalized physical activity interventions integrated into the patient's care/life trajectory
* on factors favoring adhesion to an adapted physical activity program [APA] during and/or after cancer treatment

This is a prospective, exploratory, monocentric study to explore these points.

As part of routine management in the immunohaemato-oncology [IHO] department of the Grenoble Alpes University Hospital, a personalized physical activity [PA] program is systematically proposed by a PA professional, with a program adapted to the child, his or her motivations and limitations.

As part of the protocol, a questionnaire-based assessment of motivations and obstacles, as well as quality of life, will be carried out at the start of the PA program and again after 4 to 6 months. Criteria for adherence to the APA program will also be collected.

EXPECTED OUTPUTS

* Propose an organizational model in pediatric oncology for the early and sustained practice of APA with children and adolescents hospitalized for cancer.
* Finalize assessment and follow-up materials for children receiving APA support in pediatric oncology (information leaflets, certificate of no contra-indication to APA, assessment and follow-up form, questionnaire on attitude and motivation to APA, etc.).
* Provide guidance to help young cancer patients adhere more effectively to APA program.
* Participate in the promotion of APA and the development of APA recommendations for children and adolescents treated for cancer, in conjunction with the SFCE (Children Cancer French Society) national working group on APA for children and adolescents with cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 3 years to under 18 years under care at Grenoble Alpes University Hospital
* New cancer diagnosis or relapse in the absence of previous APA treatment
* All cancer pathologies:

Diagnosis of acute or chronic hematological malignancy OR Central nervous system tumors OR Other solid tumors

* Regardless of therapeutic pathway
* Parents and patient over 5 years old understanding french langage
* Patient and parents who have not objected to participation after being informed

Exclusion Criteria:

* Patient with a strict medical contraindication to physical activity identified by the referring physician or another specialist physician, particularly the sports physician (unstabilized heart or lung disease, uncontrolled diabetes, etc.)

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children with cancer taken in charge in the paediatric immuno haematology service of the Grenoble Alpes University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 48 (Estimated)
Dates: Start 2024-02-16 (Actual); Primary Completion 2025-08-16 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Adhesion to an APA programm | 4 to 6 months
  Adherence of children and adolescents undergoing cancer treatment to personalized support in Adapted Physical Activity [APA] offered at an early stage and for a minimum duration of 4 to 6 months : patients following the whole APA program/patients included, in percent

SECONDARY OUTCOMES:
Motivation and restraints | 4 to 6 months
  This outcome is measured through a semi directive questionnaire elaborated by the SENS laboratory (Laboratory of physical exercice and social environment, Grenoble, France). It measures attitudes and motivations that have been identified as key factors in behavior change, within the framework of the main health psychology models of behavior change, such as the theory of planned behavior, the health action process approach, or self-determination theory .In order to measure these constructs, tools adapted to children from 8 years old and scientifically validated were identified in the scientific literature and adapted for the APADHOP project.
  Children with cancer over 8 years old and one or both parents will answer to questions at the start of the adapted physical activity programm ((APA) and after 4 to 6 months of APA personnalised support.
  There is no scoring as this is a descriptive outcome (after been analyzed by a humanities and social sciences researcher)
Quality of life measure | 4 to 6 months
  Quality of life will be measured by international validated PedsQL questionnaires V4.0 (paediatric quality of Life Inventory) according to the age of the patient:
  * For parents of children aged 2-4 years:
  * For parents of children aged 5 to 7
  * For parents of children aged 8 to 12
  * For parents of children aged 13 to 18
  * For children aged 5 to 7
  * For children aged 8 to 12
  * For children aged 13 to 18 This questionnaires will be administrated at the start of the adapted physical activity (APA) programm and after 4 to 6 months of personalized APA support.
  Each item of the questionnaire is scored between 0 and 4 and the total score of the questionnaire is between 0 an 100. The higher score means a better quality of life.
  To be able to measure the score at least 50% of the items must be answered. The results will be analysed only for patients and parents who have answered to the questionnaires at both evaluation time.
Representation of physical activity | 4 to 6 months
  The evaluation of the representation of physical activity Activity of children and parents at diagnosis and after 4 to 6 months of personalized APA support will be performed through a semi directive questionnaire elaborated by the SENS Laboratory (Laboratory of physical exercice and social environment, Grenoble University in France).
  The questionnaires will be administred to patients over 8 years and parents at the start of the adapted physical activity (APA) programm and after 4 to 6 months of personalized APA support. The effect of personalized support will also be studied by carrying out pre/post analyzes of these dimensions.
  There is no scoring as this is a descriptive outcome that will be analysed by humanities and social siences university researchers.

CONTACTS AND LOCATIONS:
Overall Officials: Leila Gofti Laroche, MD, Principal Investigator — CHU Grenoble Alpes
Locations (1):
- CHU Grenoble Alpes, Grenoble, Isere, France

IPD SHARING:
Plan to Share IPD: No
No individual participant data sharing